CLINICAL TRIAL: NCT00318786
Title: Trial to Investigate the Efficacy and the Safety of Thrice-Daily NN2000-Mix70 (NovoRapid 70 Mix) Compared to Twice-Daily NN-X14Mix30 (NovoRapid 30 Mix) in Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Three Times a Day BIAsp-70 Compared to Two Times a Day BIAsp-30 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1598; JapicCTI-060241 (Registry Identifier: japic)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart

SUMMARY:
This trial is conducted in Japan. This a clinical trial to study the efficacy and safety of three times a day BIAsp-70 compared to two times a day BIAsp-30 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* Current treatment using intermediate-acting, long-acting insulin (including long-acting insulin analogue) or pre-mixed human insulin for at least 24 weeks
* HbA1c at least 7.5% and below 10.0%

Exclusion Criteria:

* Proliferative retinopathy or maculopathy requiring acute treatment
* Impaired hepatic and/or renal function
* Cardiac diseases
* Uncontrolled hypertension
* Known hypoglycemia unawareness or recurrent major hypoglycemia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2006-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C (HbA1C) | After 16 weeks of treatment

SECONDARY OUTCOMES:
HbA1C, after 28 weeks of treatment; Plasma glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Kadowaki T, Nishida T, Kaku K. 28-week, randomized, multicenter, open-label, parallel-group phase III trial to investigate the efficacy and safety of biphasic insulin aspart 70 thrice-daily injections vs twice-daily injections of biphasic insulin aspart 30 in patients with type 2 diabetes. J Diabetes Investig. 2010 Jun 1;1(3):103-10. doi: 10.1111/j.2040-1124.2010.00015.x. PMID 24843416
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com